CLINICAL TRIAL: NCT02636660
Title: Health-related Quality of Life and Nursing-sensitive Outcomes in Mechanically Ventilated Patients in an Intensive Care Unit
Brief Title: Health-related Quality of Life and Nursing-sensitive Outcomes in Mechanically Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)136/2011
Record Dates: First submitted 2015-11-12; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Quality of Life
Keywords: Critical care; Mechanical Ventilation; Quality of Life; Stressors; Nursing Sensitive Outcomes; Nursing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will allow us to determine the perceived Health-Related Quality of Life (HRQL) a year after ICU discharge, and compare it with HRQL measured earlier on in the process, as well as analyse the negative experiences they had while in the ICU and as a result of MV and their impact over time. It will also allow us to assess the effect of Nursing Sensitive Outcomes and ICU stressors on health-related outcomes and how they affect HRQL.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is one the most utilised therapeutic techniques within the intensive care unit (ICU). It is commonly used to support patients diagnosed with severe respiratory failure, but several complications have been documented in the literature that can appear during both the acute phase of treatment and in later phases, becoming a chronic problem in some cases. Most of these complications are related to the length of treatment, and they could affect patients' health-related quality of life (HRQL).

HRQL conceptualisation is vital for the analysis and evaluation of health-related outcomes. Knowing the patient's health perception, his wishes and motivating factors when making decisions related to his own health, as well as applying procedures to evaluate healthcare providers are essential to the definition of HRQL.

Diagnosis and treatment of illness exclusively at a biomedical level in addition to technologically advanced procedures represent a qualitative improvement in patient survival in recent decades, but they have reduced a more holistic approach to health care because they only fight against illness without promoting patient welfare.

From a more holistic perspective and in an attempt to quantify the contribution of nursing to health-related outcomes, the term "nursing-sensitive outcome" (NSO) was created. According to the National Quality Forum, those indicators that are sensitive to certain nursing interventions are measurements of the process' structure (the process itself and its outcomes) and are affected or influenced by the intervention of nurses, although the responsibility is shared with other professionals. The forum agreed on several NSO standards such as pressure ulcer care, infection control, falls prevention, expertise of the nursing team, patient satisfaction and HRQL.

Outcome evaluation and knowledge of HRQL in mechanically ventilated critical care patients is vital to understanding how this therapeutic technique affects patients and therefore to designing care strategies for both acute and later phases of treatment. The goal is to minimize unwanted effects and improve cost-effectiveness, always considering the patient's perspective during the decision-making process.

The analysis of factors that determine the patient's perception on HRQL during the different phases of illness as well as the adaptation process to unwanted results will give us in-depth knowledge of the mechanisms that affect their HRQL in a negative way and therefore plan interventions to promote the optimal patient welfare.

There is a great deal of published literature on mechanically ventilated patient's HRQL. All authors agree that the quality of life perceived by these patients is worse than that perceived by the reference population, although the determinants of the HRQL are not well defined. Additionally, differences among critical care units (surgical, cardiac, general) and the variety of tools utilised to measure HRQL make it hard to compare results.

Highly specialised ICUs constitute a very stressful environment for the patient, which has been related to the onset of delirium or an acute confusional state in the phases of the disease , but other mid and long-term repercussions such as memory loss, delusion and other neurophysiological disturbances that have an effect on HRQL perception have been described.

Some authors have studied factors that have a stressful effect on mechanically ventilated patients and have found that one of the worst remembered and most stressful experiences, aside from thirst and pain, is endotracheal tube discomfort.

There are several tools to assess stressors within ICU, and all of them allow us to assess the degree of stress or nuisance experienced by the patient for each factor. One of the most well-known is the Intensive Care Unit Environmental Stressor Scale (ICUESS), which allows us to perform a global evaluation of the ICU but does not take into account problems secondary to tracheal intubation or MV. Another tool recently described in a HRQL study on mechanically ventilated patients is the ICU Stressful Experience Questionnaire (ICU-SEQ), which evaluates the general aspects of an ICU setting but also emphasizes those problems that originated as a result of orotracheal intubation and MV.

Knowing what HRQL is, its stressors and which NSO have an influence on it should allow us to design and implement strategies and nursing care plans to minimise negative effects and address chronic problems, thereby improving the patient's welfare, security and quality of life.

Setting The study will be carried out at the Intensive Care Unit of the Hospital Universitari Vall d'Hebron, located in Barcelona, Spain, which is a high-complexity hospital and a referral centre for many disease processes at a national level.

Sample size According to data previously collected in our department, a total of 360 patients will meet the inclusion criteria during the study timeframe. Assuming possible losses and a high mortality rate within critical care, the final cohort is expected to be 200 patients.

Sampling technique A non-probabilistic convenience sampling will be used, including patients as they are admitted to the ICU.

Variables The following variables will be collected: anthropometric and sociodemographic data and data related to ICU admission, mechanical ventilation, NSO, HRQL and ICU stressors.

Assessment Tools To assess HRQL, the Short-Form-36 Health Survey (SF-36) will be used. For a more specific assessment on respiratory issues, the Saint Georges Respiratory Questionnaire (SGRQ) will be used. Both questionnaires have been validated in Spanish.

To evaluate ICU stressors, the ICU Stressful Experience Questionnaire (ICU-SEQ) will be used. This tool was created by Rotondi and modified by Samuelson. In addition to evaluating general ICU experiences, it also evaluates experiences related to the endotracheal tube.

To translate and adapt the ICU-SEQ into Spanish, the following process will be used:

1. Translation and back translation into Spanish by two bilingual translators.
2. Transcultural adaptation via a pilot study to assess proper comprehension of the different items.

Data Collection Data will be collected over 12 consecutive months. Patient selection for the study cohort will be performed by the research team by evaluating all patients who may need or had needed MV. Follow up documentation will be provided for all mechanically ventilated patients. When a patient has been mechanically ventilated for over 48 hours, informed consent will be obtained from the next of kin. From that moment, all patient data from their medical records will be gathered until MV is discontinued.

One week after the patient has been discharged from the ICU, informed consent will be obtained from the patient. Approaching the patient earlier is considered to be inappropriate by the research team. If the patient agrees to participate in the study, the SF-36, SGRQ and ICU-SEQ questionnaires will be provided for the patient to complete. The same questionnaires will be given to the main caregiver at that time.

One year after ICU discharge, the same questionnaires will be completed again by the patient to assess the persistency of stressors' sequelae.

Data Analysis A descriptive analysis will be carried out for all variables. Mean and standard deviation will be utilised for quantitative variables that follow a normal distribution. For the rest of the variables, the median, maximum and minimum values will be used. Qualitative variables will be described utilising absolute frequencies and percentage values for each category.

Statistical analysis of HRQL results will be performed on the questionnaire's different dimensions as well as on the questionnaire as a whole. To compare the results obtained at the time of ICU discharge with those obtained one year after discharge, Student's t-test or Wilcoxon test will be applied to the paired data depending on the variable distribution. This analysis will also depend on the length of MV.

A multiple regression model will be elaborated utilising as HRQL as the result variable. Relevant clinical situations (number of transfusions and surgical interventions, pressure ulcers, nosocomial infections…) will be considered as independent variables.

All analysis will be performed with a 95% confidence interval.

Limitations and Bias The main limitation of this study is that the patient's quality of life one year after ICU discharge could be affected by non-identifiable events that have no relation to those studied. The main bias is the patient's memory because the patients will be asked about events that may be difficult to recall.

Ethical considerations This study has been approved by the Ethics Committee of Clinical Investigation of the Hospital Universitari Vall d'Hebron.

Informed consent will be obtained from patients and main caregivers, always making sure participants' confidentiality and anonymity is preserved through the process.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Mechanical ventilation for more than 48 hours.
* Voluntary participation (signed informed consent).

Exclusion Criteria:

* Patients admitted from other ICUs that had been mechanically ventilated for more than 48 hours at the time of admission to our centre.
* Patients with domiciliary respiratory support.
* Mentally or psychologically impaired patients (unable to comprehend the questionnaire).
* Patients who do not speak Spanish fluently.
* Patient without a permanent address (unable to do a proper follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All mechanically ventilated patients admitted to our intensive care unit that fulfill the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQL) of patients admitted to ICU | 2 weeks after discharge from ICU
Health-Related Quality of Life (HRQL) of patients admitted to ICU | 1 year after discharge for ICU

SECONDARY OUTCOMES:
Differences in HRQL in mechanically ventilated patients prior to admission into ICU and one year after discharge from the ICU | 1 year after discharge for ICU
Relationship between the duration (in days) of mechanical ventilation and HRQL one year after discharge from the ICU | 1 year after discharge for ICU
Relationship between Nursing Sensitive Outcome 1 (Pressure Ulcer Care) and the HRQL of mechanically ventilated patients in ICU. | 1 year after discharge for ICU
  Number and location of pressure ulcers
Relationship between Nursing Sensitive Outcome 2 (Falls Prevention) and the HRQL of mechanically ventilated patients in ICU. | 1 year after discharge for ICU
  Numbers of unintentional falls
Relationship between Nursing Sensitive Outcome 3 (Infection Control) and the HRQL of mechanically ventilated patients in ICU. | 1 year after discharge for ICU
  number of nosocomial infections: urinary tract infections, tracheobronquitis and CVC-related infections
Relationship between Nursing Sensitive Outcome 4 (Expertise of the Nursing Team) and the HRQL of mechanically ventilated patients in ICU. | 1 year after discharge for ICU
  measured in 3 intervals: less than 1 year, between 1 and 5 years, and more than 5 years experience in ICU
Differences between the patient's own assessment of HRQL and the main caregiver's perception. | 1 year after discharge for ICU
Number of stressors that mechanically ventilated patients admitted in ICU identify when discharged utilizing the ICU Stressful Experience Questionnaire (ICU-SEQ) | 1 year after discharge for ICU
Relationship between the amount and type of stressors perceived by mechanically ventilated patients during their admission and their HRQL one year after discharge from the ICU | 1 year after discharge for ICU

CONTACTS AND LOCATIONS:
Overall Officials: Maria Alba Riera Badia, Principal Investigator — Nursing Supervisor

REFERENCES:
- [Result] Frutos F, Allía I, Lorenzo MR, García PArdo J, Nolla M et al. Utilización de la ventilación mecánica en 72 unidades de cuidados intensivos en España. Medicina Intensiva 2003;27(1):1-12.
- [Result] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Result] Dowdy DW, Eid MP, Dennison CR, Mendez-Tellez PA, Herridge MS, Guallar E, Pronovost PJ, Needham DM. Quality of life after acute respiratory distress syndrome: a meta-analysis. Intensive Care Med. 2006 Aug;32(8):1115-24. doi: 10.1007/s00134-006-0217-3. Epub 2006 Jun 17. PMID 16783553
- [Result] Combes A, Costa MA, Trouillet JL, Baudot J, Mokhtari M, Gibert C, Chastre J. Morbidity, mortality, and quality-of-life outcomes of patients requiring >or=14 days of mechanical ventilation. Crit Care Med. 2003 May;31(5):1373-81. doi: 10.1097/01.CCM.0000065188.87029.C3. PMID 12771605
- [Result] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Result] Schwartzmann L. Calidad de vida relacionada con la salud: aspectos conceptuales. Ciencia y enfermería 2003;IX(2):9-21.
- [Result] Chatila W, Kreimer DT, Criner GJ. Quality of life in survivors of prolonged mechanical ventilatory support. Crit Care Med. 2001 Apr;29(4):737-42. doi: 10.1097/00003246-200104000-00007. PMID 11373458
- [Result] Chelluri L, Im KA, Belle SH, Schulz R, Rotondi AJ, Donahoe MP, Sirio CA, Mendelsohn AB, Pinsky MR. Long-term mortality and quality of life after prolonged mechanical ventilation. Crit Care Med. 2004 Jan;32(1):61-9. doi: 10.1097/01.CCM.0000098029.65347.F9. PMID 14707560
- [Result] McKinley S, Fien M, Elliott R, Elliott D. Health-Related Quality of Life and Associated Factors in Intensive Care Unit Survivors 6 Months After Discharge. Am J Crit Care. 2016 Jan;25(1):52-8. doi: 10.4037/ajcc2016995. PMID 26724295
- [Result] Douglas SL, Daly BJ, Gordon N, Brennan PF. Survival and quality of life: short-term versus long-term ventilator patients. Crit Care Med. 2002 Dec;30(12):2655-62. doi: 10.1097/00003246-200212000-00008. PMID 12483055
- [Result] Novaes MA, Knobel E, Bork AM, Pavao OF, Nogueira-Martins LA, Ferraz MB. Stressors in ICU: perception of the patient, relatives and health care team. Intensive Care Med. 1999 Dec;25(12):1421-6. doi: 10.1007/s001340051091. PMID 10660851
- [Result] Granja C, Lopes A, Moreira S, Dias C, Costa-Pereira A, Carneiro A; JMIP Study Group. Patients' recollections of experiences in the intensive care unit may affect their quality of life. Crit Care. 2005 Apr;9(2):R96-109. doi: 10.1186/cc3026. Epub 2005 Jan 31. PMID 15774056
- [Result] Roberts BL, Rickard CM, Rajbhandari D, Reynolds P. Factual memories of ICU: recall at two years post-discharge and comparison with delirium status during ICU admission--a multicentre cohort study. J Clin Nurs. 2007 Sep;16(9):1669-77. doi: 10.1111/j.1365-2702.2006.01588.x. PMID 17727586
- [Result] Rotondi AJ, Chelluri L, Sirio C, Mendelsohn A, Schulz R, Belle S, Im K, Donahoe M, Pinsky MR. Patients' recollections of stressful experiences while receiving prolonged mechanical ventilation in an intensive care unit. Crit Care Med. 2002 Apr;30(4):746-52. doi: 10.1097/00003246-200204000-00004. PMID 11940739
- [Result] Samuelson KA. Unpleasant and pleasant memories of intensive care in adult mechanically ventilated patients--findings from 250 interviews. Intensive Crit Care Nurs. 2011 Apr;27(2):76-84. doi: 10.1016/j.iccn.2011.01.003. Epub 2011 Mar 2. PMID 21371888
- [Result] Tembo A, Parker V, Higgins I. The lived experience of critically ill patients in intensive care - A phenomenological inquiry. Australian Critical Care 2013;26(2):82.
- [Result] Mendelsohn AB, Chelluri L. Interviews with intensive care unit survivors: assessing post-intensive care quality of life and patients' preferences regarding intensive care and mechanical ventilation. Crit Care Med. 2003 May;31(5 Suppl):S400-6. doi: 10.1097/01.CCM.0000065278.90460.F0. No abstract available. PMID 12771591
- [Result] Tsay SF, Mu PF, Lin S, Wang KW, Chen YC. The experiences of adult ventilator-dependent patients: a meta-synthesis review. Nurs Health Sci. 2013 Dec;15(4):525-33. doi: 10.1111/nhs.12049. Epub 2013 Mar 11. PMID 23480454
- [Result] Azoulay E, Kentish-Barnes N, Pochard F. Health-related quality of life: an outcome variable in critical care survivors. Chest. 2008 Feb;133(2):339-41. doi: 10.1378/chest.07-2547. No abstract available. PMID 18252911
- [Derived] Riera A, Gallart E, Vicalvaro A, Lolo M, Solsona A, Mont A, Gomez J, Tellez D, Fuentelsaz-Gallego C. Health-related quality of life and nursing-sensitive outcomes in mechanically ventilated patients in an Intensive Care Unit: a study protocol. BMC Nurs. 2016 Feb 5;15:8. doi: 10.1186/s12912-016-0127-9. eCollection 2016. PMID 26855613